CLINICAL TRIAL: NCT02637076
Title: Does Xyrem Influence Brain Dopamine in Patients With Narcolepsy? A PET Imaging Investigation
Brief Title: Xyrem and Brain Dopamine in Narcolepsy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Responsible Party: Principal Investigator, Stephen Kish, Senior Scientist, Head Human Brain Lab, Centre for Addiction and Mental Health
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 017-2014
Record Dates: First submitted 2015-12-17; First posted 2015-12-22 (Estimated); Results first posted 2021-03-23 (Actual); Last update posted 2021-03-23 (Actual); Status verified 2021-02

CONDITIONS: Narcolepsy With Cataplexy; Healthy Controls
Keywords: Xyrem; narcolepsy with cataplexy; positron emission tomography; dopamine
MeSH Terms: conditions — Narcolepsy | interventions — Sodium Oxybate

STUDY DESIGN:
Intervention Model Description: Participants will be recruited to fill 2 separate study groups: 1) participants with a diagnosis of narcolepsy with cataplexy; 2) healthy controls.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- narcolepsy with cataplexy (Experimental): patients given single dose of Xyrem
  Interventions: Drug: Xyrem
- healthy controls (Experimental): healthy controls given a single dose of Xyrem
  Interventions: Drug: Xyrem

INTERVENTIONS:
Drug: Xyrem — single 3.0 gram dose
  Other Names: Sodium Oxybate; gamma-hydroxybutyrate

SUMMARY:
The overall aim of this investigation is to establish whether an action of Xyrem® on the brain dopamine system in patients with narcolepsy, and in a comparison control group, might explain part of the anti-narcoleptic effect of the drug.

Trial Objective is to establish, using positron emission tomography (PET), in Xyrem®-naïve narcolepsy with cataplexy patients, and in matched controls, whether a single dose of Xyrem® causes changes in striatal binding of 11C-raclopride and 11C-DTBZ that would suggest altered activity of brain dopamine neurones.

ELIGIBILITY:
Inclusion Criteria:

* current diagnosis of narcolepsy with cataplexy OR healthy control

Exclusion Criteria:

* use of any sedative hypnotics, tranquilizers, anticonvulsants, antihistamines (except non-sedating), benzodiazepines, clonidine or any medication known to affect dopamine at start of baseline period
* significant unstable or uncontrolled medical/psychiatric disease
* significant history of head trauma/surgery or seizure disorder
* radiation exposure exceeding 20mSv in last 12 months
* pregnancy
* substance abuse/dependence (including alcohol)
* have sleep apnea, or are shift workers
* on a sodium-restricted diet
* has ever taken Xyrem / sodium oxybate / GHB at any time
* claustrophobia
* metal implants / objects in the body that may interfere with MRI
* succinic semialdehyde dehydrogenase deficiency

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2016-01; Primary Completion 2020-01-23 (Actual); Study Completion 2020-01-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen J Kish, Ph.D., Principal Investigator — Centre for Addiction and Mental Health
Locations (1):
- Centre for Addiction and Mental Health (CAMH), Toronto, Ontario, Canada

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Narcolepsy With Cataplexy | Healthy Controls
Started | 2 | 15
Completed | 1 | 10
Not Completed | 1 | 5
Not completed — due to technical difficulties, the 1 hour post PET scan was not completed at the one hour time point | 1 | 1
Not completed — Withdrawal by Subject | 0 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Narcolepsy With Cataplexy | Healthy Controls | Total
Number analyzed (Participants) | 1 | 10 | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 52 | 29.6 (8) | 31.6 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 4 | 5
  Male | 0 | 6 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 1 | 10 | 11
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 6 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 1 | 3 | 4
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 1 | 10 | 11
[C-11]raclopride BPND at Baseline [Mean (Standard Deviation); unit: BPND (Binding Potential)] — [C-11] raclopride is a radioligand that binds to the D2/3 dopamine receptor in the dopamine-rich striatum and which is sensitive to dopamine occupancy.
  BPND (Binding Potential)
    Limbic Striatum | 2.59 | 2.83 (0.19) | 2.80 (0.19)
    Associative Striatum | 3.06 | 3.63 (0.32) | 3.58 (0.35)
    Sensorimotor Striatum | 3.11 | 4.04 (0.43) | 3.96 (0.49)
[C-11]DTBZ BPND at Baseline [Mean (Standard Deviation); unit: BPND (Binding Potential)] — [C-11] DTBZ is a radioligand that binds to the vesicular monoamine transporter and which is sensitive to dopamine occupancy.
  BPND (Binding Potential)
    Limbic Striatum | 1.68 | 1.85 (0.19) | 1.84 (0.18)
    Associative Striatum | 2.41 | 2.60 (0.26) | 2.58 (0.25)
    Sensorimotor Striatum | 2.49 | 3.05 (0.38) | 3.00 (0.40)

OUTCOME MEASURES:

1. Primary Outcome: [C-11]Raclopride BPND at 1 Hour Post Xyrem
Description: BPND (Binding Potential) of [C-11]raclopride measures 1 hour after taking a single 3g dose of Xyrem.
Time Frame: 1 hour post Xyrem
Measure: Mean (Standard Deviation); unit: BPND (Binding Potential)
Arm/Group | Narcolepsy With Cataplexy | Healthy Controls
Number analyzed (Participants) | 1 | 10
BPND (Binding Potential)
  Limbic Striatum | 2.94 | 3.01 (0.28)
  Associate Striatum | 3.80 | 3.70 (0.33)
  Sensorimotor Striatum | 3.87 | 4.11 (0.49)
Statistical Analysis 1: Comparison: Healthy Controls; Test type: Other; p = 0.31, repeated measures ANOVA; F(2,36)=1.26

2. Primary Outcome: % Change in PET [C11]Raclopride Binding From Baseline After Single Dose of Xyrem
Description: [C-11] raclopride is a radioligand that binds to the D2/3 dopamine receptor in the dopamine-rich striatum and which is sensitive to dopamine occupancy.
  % change was calculated as follows: (1 hour BPND - baseline BPND)/baseline BPND *100; Mean % change represents the mean of each participant's individual % change within the group.
Time Frame: 1 hour post Xyrem
Measure: Mean (Standard Deviation); unit: percentage change from baseline
Arm/Group | Narcolepsy With Cataplexy | Healthy Controls
Number analyzed (Participants) | 1 | 10
percentage change from baseline
  Limbic Stiatum | 13.27 | 6.49 (8.60)
  Associative Striatum | 23.88 | 2.11 (8.59)
  Sensorimotor Striatum | 24.43 | 1.93 (8.85)

3. Primary Outcome: [C-11]Raclopride BPND at 7 Hours Post Xyrem
Description: BPND (Binding Potential) of [C-11]raclopride measures 7 hours after taking a single 3g dose of Xyrem.
Time Frame: 7 hours post Xyrem
Measure: Mean (Standard Deviation); unit: BPND (Binding Potential)
Arm/Group | Narcolepsy With Cataplexy | Healthy Controls
Number analyzed (Participants) | 1 | 10
BPND (Binding Potential)
  Limbic Striatum | 2.33 | 2.76 (0.18)
  Associate Striatum | 2.83 | 3.62 (0.29)
  Sensorimotor Striatum | 2.75 | 4.06 (0.40)

4. Primary Outcome: % Change in PET [C11]Raclopride Binding From Baseline After Single Dose of Xyrem
Description: [C-11] raclopride is a radioligand that binds to the D2/3 dopamine receptor in the dopamine-rich striatum and which is sensitive to dopamine occupancy.
  % change was calculated as follows: (7 hours BPND - baseline BPND)/baseline BPND *100; Mean % change represents the mean of each participant's individual % change within the group.
Time Frame: 7 hours post Xyrem
Measure: Mean (Standard Deviation); unit: percentage change from baseline
Arm/Group | Narcolepsy With Cataplexy | Healthy Controls
Number analyzed (Participants) | 1 | 10
percentage change from baseline
  Limbic Striatum | -10.13 | -2.07 (8.24)
  Associative Striatum | -7.50 | 0.17 (7.42)
  Sensorimotor Striatum | -11.56 | 0.72 (7.64)

5. Secondary Outcome: [C-11]DTBZ BPND at 5 Hours Post Xyrem
Description: Measurement of [C-11]DTBZ 5 hours after taking a single dose of 3g Xyrem
Time Frame: 5 hours post single Xyrem dose
Measure: Mean (Standard Deviation); unit: BPND (binding potential)
Arm/Group | Narcolepsy With Cataplexy | Healthy Controls
Number analyzed (Participants) | 1 | 10
BPND (binding potential)
  Limbic Striatum | 1.71 | 1.82 (0.24)
  Associative Striatum | 2.56 | 2.65 (0.40)
  Sensorimotor Striatum | 2.65 | 3.12 (0.53)

6. Secondary Outcome: % Change in PET [C-11] Dihydrotetrabenazine (DTBZ) Binding From Baseline to Five Hours Post Xyrem
Description: [C-11] DTBZ is a radioligand that binds to the vesicular monoamine transporter and which is sensitive to dopamine occupancy.
  % change was calculated as follows: (5 hour BPND - baseline BPND)/baseline BPND *100; Mean % change represents the mean of each participant's individual % change within the group.
Time Frame: 5 hours post single Xyrem dose
Measure: Mean (Standard Deviation); unit: percentage change from baseline
Arm/Group | Narcolepsy With Cataplexy | Healthy Controls
Number analyzed (Participants) | 1 | 10
percentage change from baseline
  Limbic Striatum | 2.00 | -1.98 (9.20)
  Associative Striatum | 6.10 | 2.04 (11.84)
  Sensorimotor Striatum | 6.51 | 2.47 (12.09)
Statistical Analysis 1: Comparison: Healthy Controls; Test type: Other; p = 0.748, repeated measures ANOVA

7. Secondary Outcome: Blood Gamma-hydroxybutyrate (GHB) Concentration (AUC)
Description: The concentration of gammahydroxybutyrate in blood of participants who have received a single dose of Xyrem, as measured by Area Under the Curve.
Time Frame: multiple time points from 0 to 7 hours post-Xyrem
Measure: Mean (Standard Deviation); unit: AUC (ug/ml*hr)
Arm/Group | Narcolepsy With Cataplexy | Healthy Controls
Number analyzed (Participants) | 1 | 10
AUC (ug/ml*hr) | 187.03 | 178.49 (52.12)

8. Secondary Outcome: Blood Gamma-hydroxybutyrate (GHB) Cmax
Description: The concentration of gammahydroxybutyrate in blood of participants who have received a single dose of Xyrem as measured by Cmax.
Time Frame: multiple time points from 0 to 7 hours post-Xyrem
Measure: Mean (Standard Deviation); unit: mg/ml
Arm/Group | Narcolepsy With Cataplexy | Healthy Controls
Number analyzed (Participants) | 1 | 10
mg/ml | 107 | 107.37 (32.95)

9. Secondary Outcome: Duration of Drowsiness
Description: Period of time when the participant was experiencing the sedative action of Xyrem. Data derived from self-report as well as anesthesiologist observation.
Time Frame: observed after receiving single dose of Xyrem, up to 9 hours
Measure: Median (Full Range); unit: minutes
Arm/Group | Narcolepsy With Cataplexy | Healthy Controls
Number analyzed (Participants) | 1 | 10
minutes | 220.20 | 92.4 [10.02 to 285.00]

ADVERSE EVENTS:
Time Frame: Adverse events will be assessed at each study visit following administration of the first PET radiotracer until the follow-up phone after Xyrem administration (2 visits plus 1 follow-up phone call), an average of 10 days per participant.
Arm/Group | Narcolepsy With Cataplexy | Healthy Controls
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/15
Other Adverse Events (participants affected / at risk) | 0/2 | 4/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Narcolepsy With Cataplexy (N=2) | Healthy Controls (N=15)
Euphoria (General disorders) | 0 (0) | 1 (1)
Nausea (General disorders) | 0 (0) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-09-13): https://cdn.clinicaltrials.gov/large-docs/76/NCT02637076/Prot_SAP_000.pdf
  • Informed Consent Form (2019-02-27): https://cdn.clinicaltrials.gov/large-docs/76/NCT02637076/ICF_001.pdf